CLINICAL TRIAL: NCT07098013
Title: Adherence and Efficacy of an Unguided Internet-Based Relaxation Program for Stress and Anxiety: Insights From Two Randomized Controlled Trials
Brief Title: Unguided Internet-based Relaxation Program for Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eotvos Lorand University (Other)
Responsible Party: Principal Investigator, Luca Csirmaz, Principal Investigator, Eotvos Lorand University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023/603; PD 143491 (Other Grant/Funding Number: National Scientific Fund)
Record Dates: First submitted 2025-07-18; First posted 2025-08-01 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Anxiety; Stress (Psychology)
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Internet-based Anxiety Intervention (Experimental): Participants received access to a fully automated, unguided internet-based relaxation program designed to reduce stress and anxiety. The program included evidence-based audio exercises such as mindfulness, deep breathing, progressive muscle relaxation, imagery, and acceptance-based practices. In Trial 1, participants completed a 4-week version with 28 short daily exercises. In Trial 2, a modified 3-week version with longer, fewer sessions. All materials were delivered in English to Hungarian non-native speakers via a website, without therapist support.
  Interventions: Behavioral: Relaxation Self-Coach
- Waitlist Control (No Intervention): Participants in the control arm were placed on a waitlist and did not receive access to the relaxation program during the active intervention phase. They were informed that they would gain full access to the same program after completing post-intervention assessments. During the waiting period, they completed the same online self-assessments (e.g., stress, anxiety, depression scales) as the intervention group. Automated reminder emails encouraged assessment completion and informed participants of their upcoming access to the program. No therapeutic content was delivered during the waitlist period.

INTERVENTIONS:
Behavioral: Relaxation Self-Coach — This intervention is a fully automated, unguided internet-based relaxation program in English. Unlike many digital mental health programs, it required no therapist involvement or incentives and was structured for real-world use. It combined evidence-based techniques-mindfulness, deep breathing, progressive muscle relaxation, guided imagery, and acceptance practices-delivered via audio modules. The program was tested in two formats: a 4-week daily format (28 sessions) and a revised 3-week modular format (21 sessions) with enhanced usability and adherence features, such as a simplified multimedia interface, reminder emails, and optional reflection prompts.
  Arms: Internet-based Anxiety Intervention

SUMMARY:
This study aimed to evaluate the effectiveness and adherence of a fully automated, unguided internet-based relaxation program designed to reduce stress and anxiety in Hungarian adults with English proficiency. Conducted through two randomized controlled trials, the program delivered evidence-based audio exercises (e.g., mindfulness, breathing, progressive muscle relaxation, and imagery techniques) via the web. The key research questions were whether this non-native English language program could reduce symptoms of anxiety, stress, and depression, and whether adherence could be improved through design modifications. The first trial tested the original 4-week version, while the second trial tested a 3-week modified version with adherence-enhancing features. Primary outcomes included changes in anxiety, depression, and stress. The study contributes to understanding the feasibility and potential of low-cost, language-accessible digital interventions for underserved populations in less structured, real-world settings.

DETAILED DESCRIPTION:
Study 1 tested a four-week program called the "28-day Relaxation Challenge." It included seven short audio sessions per week (3-12 minutes), incorporating mindfulness, mantra meditation, progressive muscle relaxation, guided imagery, acceptance-based techniques, and imaginal exposure. Participants were instructed to complete one audio session daily. Weekly assessments were administered to track engagement and symptom change. The content was housed on a Google Drive folder, and access to new exercises was contingent on completing weekly questionnaires.

Based on findings from the first trial, Study 2 implemented several design enhancements aimed at improving adherence. The revised program reduced the duration from four to three weeks and repackaged the content into fewer but longer weekly modules (3-4 per week, 9-23 minutes each), integrating several techniques into each module. Delivery was upgraded to a streamlined website interface, incorporating videos with on-screen text, simplified navigation, and built-in reminders. Motivational and reinforcement emails, as well as reflective end-of-week questions, were introduced to foster intrinsic motivation and usability. The intervention remained fully automated and unguided.

Both trials used waitlist control groups and were conducted with a 1:1 allocation ratio. Participants were recruited through Hungarian psychoeducational social media platforms without geographic or financial restrictions. Outcome measures included the Depression Anxiety Stress Scales (DASS-21), State-Trait Anxiety Inventory (STAI), and Perceived Stress Scale (PSS), among others. Adherence was monitored via self-reported engagement and weekly check-ins.

Statistical analyses included both per-protocol and modified intention-to-treat (MITT) frameworks. The MITT sample included those who completed the first weekly assessment, serving as a proxy for program initiation.

This research contributes to the understanding of how design adjustments in unguided digital mental health programs influence engagement and outcomes in real-world populations, particularly among non-native English speakers accessing interventions in English. The study also offers practical insight into feasible low-cost solutions for stress and anxiety in underserved populations.

ELIGIBILITY:
Inclusion criteria:

* being at least 18 years old
* having a self-reported at least medium level English proficiency
* Internet literacy (an an implicit eligibility criterion, as the whole procedure was done entirely online)

There was no exclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1186 (Actual)
Dates: Start 2023-06-03 (Actual); Primary Completion 2024-04-03 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
State and Trait Anxiety Inventory | Pre-and postintervention (intervention lasts 4 weeks in Trial 1, and 3 weeks in Trial 2).
  The State-Trait Anxiety Inventory consists of two 20-item subscales measuring state anxiety (temporary) and trait anxiety (general disposition). Each item is scored from 1 to 4, yielding subscale scores ranging from 20 to 80. Higher scores reflect worse anxiety levels.
Depression, Anxiety and Stress Scale | Pre- and postintervention (intervention lasts 4 weeks in Trial 1 and 3 weeks in Trial 2) + at the end of each week during treatment (at the end of week 1, week 2 and week 3 in Trial 1).
  The DASS-21 is a self-report instrument comprising three 7-item subscales measuring depression, anxiety, and stress. Each item is rated on a 4-point scale (0-3), resulting in subscale scores ranging from 0 to 21. Higher scores indicate worse symptoms (i.e., more severe depression, anxiety, or stress).
Perceived Stress Scale | Pre- and post-intervention (after 4 weeks in Trial 1, and after 3 weeks in Trial 2).
  The Perceived Stress Scale is a 10-item measure assessing perceived stress over the past month. Items are scored from 0 (never) to 4 (very often), with total scores ranging from 0 to 40. Higher scores represent worse outcomes, indicating greater perceived stress.

SECONDARY OUTCOMES:
Burnout (Maslach Burnout Inventory - General Survey) | Pre- and post-intervention. (intervention lasts 4 weeks in Trial 1, and 3 weeks in Trial 2)
  The Maslach Burnout Inventory measures burnout across three subscales: Emotional Exhaustion, Cynicism (Depersonalization), and Personal Accomplishment. Each item is rated on a 7-point scale (0-6), with higher scores on Emotional Exhaustion and Cynicism indicating worse burnout, and higher scores on Personal Accomplishment indicating a better outcome (i.e., less burnout).
Self-Efficacy (General Self-Efficacy Scale, GSE) | Pre- and post-intervention. (intervention lasts 4 weeks in Trial 1, and 3 weeks in Trial 2)
  The General Self-Efficacy Scale contains 10 items scored from 1 (not at all true) to 4 (exactly true), yielding a total score range of 10 to 40. Higher scores reflect better outcomes, indicating greater perceived self-efficacy.
Resilience (Connor-Davidson Resilience Scale, CD-RISC-10) | Pre- and post-intervention. (intervention lasts 4 weeks in Trial 1, and 3 weeks in Trial 2)
  The CD-RISC-10 assesses resilience using 10 items scored from 0 (not true at all) to 4 (true nearly all the time), with total scores ranging from 0 to 40. Higher scores indicate better resilience and psychological adaptability.

CONTACTS AND LOCATIONS:
Locations (1):
- Eötvös Loránd University PPK Psychology Department, Budapest, Hungary

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) is available to researchers upon request.
Supporting Information: Study Protocol, SAP, ICF